CLINICAL TRIAL: NCT06131788
Title: Evaluation of an Educational Hand Washing Intervention With a Single-dose Hydroalcoholic Solution on Abscesses in People Who Self-inject Drugs
Brief Title: Evaluation of an Educational Intervention on Abscesses in People Who Self-inject Drugs
Acronym: HAWA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: AIDES (Unknown); Nouvelle Aube (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: C22-61
Record Dates: First submitted 2023-10-13; First posted 2023-11-14 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-02

CONDITIONS: People Who Inject Drugs
Keywords: Harm Reduction; Soft Skin and Tissues Infections; Community-Based Participatory Research
MeSH Terms: conditions — Harm Reduction

STUDY DESIGN:
Intervention Model Description: The HAWA study is a community-based participatory research conducted in 22 harm reduction centres in France which will be cluster randomised to determine those who will propose the intervention (standard services + brief education to hand washing + MONO-RUB distribution) and those who will be the control group (standard services). After randomization, each group of HR centres will include 220 PWID within an inclusion period of 12 months and a follow-up period of 6 months.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Arm (Active Comparator): The intervention among people who inject drugs (PWID) from the intervention arm consist in : i) educational hand washing training ("fingertips first" model), ii) supply of single use alcohol-based hand rub (called MONO-RUB).
  Only staff from the 11 harm reduction (HR) centres in the intervention arm will be trained in the educational hand-washing intervention.
  Interventions: Behavioral: Educational hand hygiene intervention
- Control Arm (No Intervention): The 11 control arm HR centres will be the placebo group. People who inject drugs (PWID) in this group will receive standard HR services, including to reduce abscesses if necessary. MONO-RUBs will not be made available in these HR centres during the intervention period.

INTERVENTIONS:
Behavioral: Educational hand hygiene intervention — The intervention combines training in hand-washing with the supply of a single-use alcohol-based hand rub, called MONO-RUB
  Arms: Intervention Arm

SUMMARY:
The goal of this cluster randomised controlled trial (cRCT) is to to evaluate the effectiveness of an educational intervention combining training in hand-washing with the supply of MONO-RUBs on the reduction of skin abscesses (both observed and self-reported) in people who inject drugs (PWID).

The main questions it aims to answer are:

* does an educational intervention change the incidence of injection-related skin and soft tissue infection (SSTI) like abscesses in PWID?
* does the educational hand-washing intervention improve injection practices in terms of hand-hygiene in PWID?

According to cluster randomisation, PWID will be assigned to:

* Standard harm reduction (HR) services to reduce abscesses plus an educational hand-washing intervention (intervention arm)
* Standard HR services only (control arm)

To measure the effectiveness of the educational hand-washing intervention, the primary outcome will be the reduction in abscess prevalence compared in both groups. Statistical analyses for the primary outcome will involve comparing the reduction in abscess prevalence in the intervention arm with that in the control arm. This prevalence will be measured from observed and self-declared data, collected from the injection-site photographs and the face-to-face injection-related SSTI questionnaire, respectively.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years old,
* French-speaking,
* reporting to have injected drugs at least once during the previous week,
* and providing free and informed consent to participate.

Exclusion Criteria:

* not regularly going to the participating HR centre in the relevant city,
* having an alcohol and/or alcohol-based hand rub (ABHR) excipient intolerance/allergy,
* being under legal protection (guardianship or judicial protection),
* current pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in abscess prevalence | Month 0; Month 3; Month 6
  The primary outcome will be the change in abscess prevalence between M0 and M6, compared between the control and intervention arms, measured from observed and self-declared data, collected from the injection-site photographs and the face-to-face injection-related SSTI questionnaire, respectively

SECONDARY OUTCOMES:
Change in incidence of injection-related SSTI complications other than abscesses (e.g., cellulitis, skin ulcer, etc). | Month 0; Month 3; Month 6
  This will be assessed using the injection site photographs and the face-to-face injection-related SSTI questionnaire
Impact of the educational intervention on injection practices (use of sterile equipment, equipment sharing, and injection into a dangerous body site) | Month 0 ; Month 6
  This will be determined using data from the three computer-assisted telephon interview (CATI) questionnaires.
  The EQ-5D-5L1 questionnaire is an European quality of life scale. The first part contains questions known as the "EQ-5D descriptive system", supplemented by a visual analogue scale known as the "EQ-5D VAS". It consists of a 20 cm, graduated from 0 to 100, on which the person must indicate how he or she rates his or her current state of health, 0 being the worst possible state and and 100 being the best.
MONO RUB Compliance, tolerance and satisfaction associated with the intervention (by measuring adverse events of MONO-RUB use) | Month 6
  This will be determined by mesuring adverse events, only in the intervention arm

CONTACTS AND LOCATIONS:
Overall Officials: Perrine ROUX, PhD, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France
Locations (22):
- France (22):
  - AIDES, Angoulême
  - AIDES, Avignon
  - AIDES, Besançon
  - AIDES, Bourg-en-Bresse
  - AIDES, Chartres
  - AIDES, Clermont-Ferrand
  - AIDES, La Rochelle
  - AIDES, Laval
  - AIDES, Lille
  - AIDES, Limoges
  - AIDES, Mulhouse
  - AIDES, Nevers
  - AIDES, Niort
  - AIDES, Nîmes
  - AIDES, Paris
  - AIDES, Pau
  - AIDES, Poitiers
  - AIDES, Rennes
  - AIDES, Rouen
  - AIDES, Toulon
  - AIDES, Toulouse
  - AIDES, Tours

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through the HaWa study may be provided to qualified researchers with academic interest in harm reduction for PWID. Data or samples shared will be coded, and deidentified. Approval of the request and execution of all applicable agreements are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol, SAP
Time Frame: Data requests can be submitted starting 9 months after last article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA).

REFERENCES:
- [Background] Hrycko A, Mateu-Gelabert P, Ciervo C, Linn-Walton R, Eckhardt B. Severe bacterial infections in people who inject drugs: the role of injection-related tissue damage. Harm Reduct J. 2022 May 2;19(1):41. doi: 10.1186/s12954-022-00624-6. PMID 35501854
- [Background] Dahlman D, Hakansson A, Kral AH, Wenger L, Ball EL, Novak SP. Behavioral characteristics and injection practices associated with skin and soft tissue infections among people who inject drugs: A community-based observational study. Subst Abus. 2017 Jan-Mar;38(1):105-112. doi: 10.1080/08897077.2016.1263592. Epub 2016 Nov 29. PMID 27897966
- [Background] Sartelli M, Guirao X, Hardcastle TC, Kluger Y, Boermeester MA, Rasa K, Ansaloni L, Coccolini F, Montravers P, Abu-Zidan FM, Bartoletti M, Bassetti M, Ben-Ishay O, Biffl WL, Chiara O, Chiarugi M, Coimbra R, De Rosa FG, De Simone B, Di Saverio S, Giannella M, Gkiokas G, Khokha V, Labricciosa FM, Leppaniemi A, Litvin A, Moore EE, Negoi I, Pagani L, Peghin M, Picetti E, Pintar T, Pupelis G, Rubio-Perez I, Sakakushev B, Segovia-Lohse H, Sganga G, Shelat V, Sugrue M, Tarasconi A, Trana C, Ulrych J, Viale P, Catena F. 2018 WSES/SIS-E consensus conference: recommendations for the management of skin and soft-tissue infections. World J Emerg Surg. 2018 Dec 14;13:58. doi: 10.1186/s13017-018-0219-9. eCollection 2018. PMID 30564282
- [Background] Allegranzi B, Tartari E, Pittet D. "Seconds save lives - clean your hands": the 5 May 2021 World Health Organization SAVE LIVES: Clean Your Hands campaign. J Hosp Infect. 2021 May;111:1-3. doi: 10.1016/j.jhin.2021.03.001. Epub 2021 Mar 7. PMID 33691160
- [Background] Rosenfeld J, Berggren R, Frerichs L. A Review of the Community Health Club Literature Describing Water, Sanitation, and Hygiene Outcomes. Int J Environ Res Public Health. 2021 Feb 15;18(4):1880. doi: 10.3390/ijerph18041880. PMID 33671972
- [Background] Stein MD, Phillips KT, Herman DS, Keosaian J, Stewart C, Anderson BJ, Weinstein Z, Liebschutz J. Skin-cleaning among hospitalized people who inject drugs: a randomized controlled trial. Addiction. 2021 May;116(5):1122-1130. doi: 10.1111/add.15236. Epub 2020 Sep 21. PMID 32830383
- [Background] Phillips KT. Barriers to practicing risk reduction strategies among people who inject drugs. Addict Res Theory. 2016;24(1):62-68. doi: 10.3109/16066359.2015.1068301. Epub 2015 Jul 21. PMID 27499724
- [Background] Degenhardt L, Peacock A, Colledge S, Leung J, Grebely J, Vickerman P, Stone J, Cunningham EB, Trickey A, Dumchev K, Lynskey M, Griffiths P, Mattick RP, Hickman M, Larney S. Global prevalence of injecting drug use and sociodemographic characteristics and prevalence of HIV, HBV, and HCV in people who inject drugs: a multistage systematic review. Lancet Glob Health. 2017 Dec;5(12):e1192-e1207. doi: 10.1016/S2214-109X(17)30375-3. Epub 2017 Oct 23. PMID 29074409
- [Background] Mezaache S, Briand-Madrid L, Rahni L, Poireau J, Branchu F, Moudachirou K, Wendzinski Y, Carrieri P, Roux P. A two-component intervention to improve hand hygiene practices and promote alcohol-based hand rub use among people who inject drugs: a mixed-methods evaluation. BMC Infect Dis. 2021 Feb 25;21(1):211. doi: 10.1186/s12879-021-05895-1. PMID 33632143
- [Background] Roux P, Le Gall JM, Debrus M, Protopopescu C, Ndiaye K, Demoulin B, Lions C, Haas A, Mora M, Spire B, Suzan-Monti M, Carrieri MP. Innovative community-based educational face-to-face intervention to reduce HIV, hepatitis C virus and other blood-borne infectious risks in difficult-to-reach people who inject drugs: results from the ANRS-AERLI intervention study. Addiction. 2016 Jan;111(1):94-106. doi: 10.1111/add.13089. Epub 2015 Sep 28. PMID 26234629
- [Background] Mezaache S, Protopopescu C, Debrus M, Morel S, Mora M, Suzan-Monti M, Rojas Castro D, Carrieri P, Roux P. Changes in supervised drug-injecting practices following a community-based educational intervention: A longitudinal analysis. Drug Alcohol Depend. 2018 Nov 1;192:1-7. doi: 10.1016/j.drugalcdep.2018.07.028. Epub 2018 Sep 5. PMID 30195241
- [Background] Tschudin-Sutter S, Sepulcri D, Dangel M, Ulrich A, Frei R, Widmer AF. Simplifying the World Health Organization Protocol: 3 Steps Versus 6 Steps for Performance of Hand Hygiene in a Cluster-randomized Trial. Clin Infect Dis. 2019 Aug 1;69(4):614-620. doi: 10.1093/cid/ciy948. PMID 30395180
- [Background] Pires D, Soule H, Bellissimo-Rodrigues F, Gayet-Ageron A, Pittet D. Hand Hygiene With Alcohol-Based Hand Rub: How Long Is Long Enough? Infect Control Hosp Epidemiol. 2017 May;38(5):547-552. doi: 10.1017/ice.2017.25. Epub 2017 Mar 7. PMID 28264743
- [Derived] Balhan L, Aubert M, Lacoux C, Grau N, Levy J, Stefanowski ML, Perreaut L, Sagaon-Teyssier L, Deuffic-Burban S, Cousien A, Michels D, Costa M, Roux P. A hand-washing community-based educational intervention to reduce abscess incidence among people who inject drugs: a cluster randomised controlled clinical trial protocol (the HAWA study protocol). BMC Public Health. 2024 Oct 17;24(1):2858. doi: 10.1186/s12889-024-20299-x. PMID 39420312